CLINICAL TRIAL: NCT02945033
Title: French Prospective Randomised Double Blind Study, on Aspirin Versus Placebo in Resected Colon Cancer With PI3K Mutation
Brief Title: Study on Aspirin Versus Placebo in Resected Colon Cancer With PI3K Mutation Stage III or II High Risk
Acronym: ASPIK French
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Collaborators: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015/222/HP
Record Dates: First submitted 2016-10-20; First posted 2016-10-26 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Colorectal Cancer
Keywords: Pi3k mutation; Aspirin
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with aspirin intake (Experimental): Surgical resection of colonic adenocarcinoma stage III or II high risk will be done in accordance with local guidelines. Molecular analysis of exon 9 and 20 of PI3K will be done using operative piece. If the mutation is detected, patient with colonic adenocarcinoma stage III or II high risk will take aspirin 100 mg/day during 3 years. Blood intake will be done every 6 months to evaluate patient compliance to treatment
  Interventions: Drug: aspirin intake; Procedure: Surgical resection of colonic adenocarcinoma stage III or II high risk; Biological: Molecular analysis of exon 9 and 20 of PI3K; Biological: blood intake
- Patient with placebo intake (Placebo Comparator): Surgical resection of colonic adenocarcinoma stage III or II high risk will be done in accordance with local guidelines. Molecular analysis of exon 9 and 20 of PI3K will be done using operative piece. If the mutation is detected, patient with colonic adenocarcinoma stage III or II high risk will take placebo of aspirin 100 mg/day during 3 years. Blood intake will be done every 6 months to evaluate patient compliance to treatment
  Interventions: Drug: placebo intake; Procedure: Surgical resection of colonic adenocarcinoma stage III or II high risk; Biological: Molecular analysis of exon 9 and 20 of PI3K; Biological: blood intake

INTERVENTIONS:
Drug: aspirin intake — Patient with colonic adenocarcinoma stage III or II high risk will take aspirin 100 mg/day during 3 years
  Arms: Patient with aspirin intake
Drug: placebo intake — Patient with colonic adenocarcinoma stage III or II high risk will take placebo of aspirin 100 mg/day during 3 years
  Arms: Patient with placebo intake
Procedure: Surgical resection of colonic adenocarcinoma stage III or II high risk — Surgical resection of colonic adenocarcinoma stage III or II high risk will be done in accordance with local guidelines
Biological: Molecular analysis of exon 9 and 20 of PI3K — Molecular analysis of exon 9 and 20 of PI3K will be done using operative piece
Biological: blood intake — Blood intake will be done every 6 months to evaluate patient compliance to treatment

SUMMARY:
Four retrospective studies were recently published on efficacy of aspirin in patients with surgically resected colon cancer. Two of these studies strongly suggested that aspirin used in low doses (100 mg/d) after surgical resection of colorectal cancer with PI3K mutation could act as a targeted therapy with a major protective effect on the risk of recurrence. The other two studies did not confirm the benefit of aspirin in this situation. These four retrospective studies provide an insufficient level of evidence to demonstrate the benefit of low-dose aspirin as adjuvant to surgery for colorectal cancer. Therefore, it is necessary as recommended in the conclusion of these studies and meta-analyses to perform a randomised prospective study to validate these data.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Colonic adenocarcinoma stage III
* Colonic adenocarcinoma stage II high risk MSS:

  * T4bN0 or T4aN0 tumour penetrating the surface of the visceral peritoneum
  * or less than 12 nodes evaluated;
  * or with at least two of the following criteria:lymphatic involvement, perineural invasion, venous invasion
  * or diagnosis of bowel obstruction or perforation; or poor differentiated tumour.
* PI3K mutation, exon 9 or 20 (tumour)
* Resection R0
* WHO performance status 0-2
* Chest and abdominal CT scan ≤ 8 weeks
* Life expectancy ≥ 3 years
* Written consent signed

Exclusion Criteria:

* Anticoagulant and/or Antiaggregating treatment including clopidogrel
* Regular aspirin use (> 3 doses per week during more than 3 months the last year)
* Contraindication to Aspirin : Allergy to aspirin, Active or antecedent peptic ulcer
* Severe renal or hepatic insufficiency
* Pregnancy or nursing ongoing
* Rectal cancer
* Hereditary forms (i.e. lynch syndrome patients)
* Follow-up of the patient not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Number of patient with local or distant recurrence or second colorectal cancer or death from any cause, whichever occurred first | 3 years

SECONDARY OUTCOMES:
Number of patient with local or distant recurrence or second colorectal cancer or death from any cause, whichever occurred first | 5 years
Number of alive patient | 5 years
Number of pills taken by the patient for compliance evaluation | every 6 months during 3 years
  Number of pills taken by the patient will be assess in order to evaluate patient's compliance
Number of severe bleeding grade 3-4 events | 3 years
Number of participants with treatment-related adverse events | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MICHEL, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided